CLINICAL TRIAL: NCT05304013
Title: 10-year Follow-up of Patients With Rheumatoid Arthritis Who Received Structured Treat-to-target Therapy in Early Disease
Acronym: ARCTIC-FORWARD
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Siri Lillegraven, Senior researcher, Leader of Unit for clinical research, Diakonhjemmet Hospital
Other Study IDs: DIA2021-1/ver 1
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Long-term outcomes; Extra-articular manifestations
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA, plasma, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ARCTIC-FORWARD study is a multi-center prospective observational study investigating the long-term outcomes of rheumatoid arthritis (RA) patients who received structured treat-to-target therapy early in their disease. The main hypothesis of this project is that RA treat-to-target strategies during the first two years of disease result in beneficial long-term outcomes both with regards to joint damage, disease activity and societal costs.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is one of the most common autoimmune diseases. Recent developments in RA treatment has shown to change the outcome of RA for the early stages of the disease, with very limited loss of work participation and high rates of disease activity remission. The data on the long-term outcome for patients who received early optimal treatment is much more limited, and it is of special clinical interest to know to what extent these patients should be monitored with regards to slowly evolving joint damage, subclinical inflammation, loss of physical function and loss of work participation.

The aim of this study is to assess clinical, radiographic and functional long-term outcomes of modern RA care and to identify risk factors for progressive disease.The main hypothesis of this project is that RA treat-to-target strategies during the first two years of disease result in beneficial long-term outcomes both with regards to joint damage, disease activity and societal costs. We will perform an extensive evaluation of all patients participating in the ARCTIC study 10 years after the initiation of structured treat-to-target therapy. Outcomes include disease activity, radiographic damage, functional status, DMARD use, extra-articular manifestations including interstitial lung disease, comorbidities, survival, work participation, health care resource use, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria: All patients that entered the ARCTIC study are eligible for the follow-up study. The main inclusion criteria in the ARCTIC study were age 18-75 years, fulfilment of the 2010 ACR classification criteria for RA, DMARD naivety with indication from DMARD therapy, and symptom duration of less than two years.

Exclusion Criteria: Psychiatric or mental disorders, alcohol abuse, other substance abuse, other factors making adherence to the study protocol impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established Rheumatoid arthritis who participated in the ARCTIC trial
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Progression of radiographs joint damage | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Radiographs of hands and feet
Disease activity | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by the disease activity score (DAS)
Disease activity remission | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Remission based on disease activity score (DAS)
Physical and mental health | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by SF-36

SECONDARY OUTCOMES:
Ultrasound inflammation | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Power doppler and B-mode
Grip strength | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Measured by dynamometer
Patient reported impact of disease | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  RAID
Swollen joint count | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  44 joints
Tender joint count | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  28 joints
Tender joints | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by Ritchie Articular index
Comorbidities | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Questionnaire
C-reactive protein (CRP) | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Blood test
Erythrocyte sedimentation rate (ESR) | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Blood test
Presence of rheumatoid noduli | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Skin examination
Osteoporosis | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by Dual-energy X-ray absorptiometry (DEXA)
Medication use | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Record of disease modifying drugs antirheumatic drugs including corticosteroids
Patient global assessment of disease activity | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  0-100 visual analogue scale (VAS), with higher scores Indicating more disease activity
Physician global assessment of disease activity | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  0-100 visual analogue scale (VAS), with higher scores Indicating more disease activity
Interstitial lung disease | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by HRCT
Physical activity level | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by accelerometer
Patient reported Physical function | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by HAQ-PROMIS
Health-related quality of life | 10 At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Assessed by EQ-5D
Work Productivity | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Work Productivity and Activity Impairment Questionnaire: WPAI:RA
Pulmonary function | At the ARCTIC-FORWARD examination (10 years after initial inclusion into the ARCTIC study)
  Spirometry and DLCO

CONTACTS AND LOCATIONS:
Overall Officials: Siri Lillegraven, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (11):
- Norway (11):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital, Drammen
  - Haugesund Hospital, Helse Fonna, Haugesund
  - Sørlandet Hospital, Kristiansand
  - Revmatolog Anne Lindtner Noraas, Kristiansand
  - Østfold Hospital, Moss
  - Diakonhjemmet Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs hospital (Trondheim University hospital), Trondheim
  - Martina Hansens Hospital, Viken